## **Title Page**

**Protocol Title:** A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of MT10109L (NivobotulinumtoxinA) for the Treatment of Glabellar Lines

Protocol Number: MT10109L-001

Amendment Number: Amendment 4

**Product:** MT10109L (NivobotulinumtoxinA)

**Brief Protocol Title:** MT10109L in the Treatment of Glabellar Lines

**Development Phase: 3** 

**Sponsor Name and Legal Registered Address:** 

Allergan Sales LLC

Regulatory Agency Identifying Numbers: IND Number 121473;

EudraCT Number 2014-005300-16



| Sponsor Sign | natory: | |
|--------------|---------|---|
| | | 1 |



**Protocol Amendment Summary of Changes Table** 

| DOCUMENT HISTORY | |
|-------------------|----------------|
| Document | Date |
| Amendment 4 | September 2020 |
| Amendment 3 | February 2019 |
| Amendment 2 | November 2018 |
| Amendment 1 | September 2018 |
| Original Protocol | May 2018 |

### Amendment 4 (September 2020)

This amendment is considered to be nonsubstantial based on the criteria set forth in Article 10(a) of Directive 2001/20/EC of the European Parliament and the Council of the European Union because it neither significantly impacts the safety or physical/mental integrity of participants nor the scientific value of the study.

### **Overall Rationale for the Amendment:**

The overall rationale of this protocol amendment was to integrate feedback and recommendations from a health authority.

| Section No. and Name | Description of Change | Brief Rationale |
|---|---|---|
| Title Page | Updated sponsor signatory | Administrative |
| 11 References | Added references | References added to Section 9.4.1.2 |

## **Table of Contents**

| Title Pa | Title Page |
|---|---|
| List of 7 | f Contents3Tables6Figures6 |
| <b>1.</b> 1.1 | Protocol Summary 7 Synopsis 7 |
| 2.<br>2.1<br>2.2<br>2.3 | Introduction14Study Rationale14Background14Benefit/Risk Assessment15 |
| 3. | Objectives and Endpoints |
| <b>4.</b> 4.1 4.1.1 | Study Design19Overall Design19Clinical Hypotheses20 |
| 4.4 | End of Study Definition 21 |
| <b>5.</b> 5.1 5.2 | Study Population22Inclusion Criteria22Exclusion Criteria23 |
| 5.3<br>5.4 | Lifestyle Considerations 25 Screen Failures 26 |
| 6. | Study Intervention |
| 6.1.2<br>6.2 | Instructions for Use and Administration 28 Preparation/Handling/Storage/Accountability 29 |
| 6.4 | Study Intervention Compliance 31 Concomitant Therapy 31 |
| 652 | Passua Madigina |

| 6.6 | Dose Modification | 32 |
|---|---|---|
| 7. | Discontinuation of Study Intervention and Participant | |
| | Discontinuation/Withdrawal | |
| 7.1 | Discontinuation of Study Intervention. | |
| 7.2 | Participant Discontinuation/Withdrawal from the Study | |
| 7.3 | Lost to Follow Up | |
| <b>8.</b> | Study Assessments and Procedures | |
| 8.1<br>8.1.1 | Efficacy Assessments Facial Wrinkle Scale With Photonumeric Guide (FWS) | |
| 0.1.1 | Tueld Willikie Sedie Will I notonamene Guide (1 WS) | |
| 8.2 | Safety Assessments | 38 |
| 8.2.1 | Adverse Events | 38 |
| 8.2.2 | Physical Examination | 38 |
| 8.2.4 | Vital Signs | |
| 8.2.5 | Electrocardiograms | |
| 8.2.6 | Hematology and Blood Chemistry | |
| 8.2.7 | Urine Pregnancy Tests | 40 |
| 8.2.8 | Suicidal Risk Monitoring. | |
| 8.3 | Adverse Events and Serious Adverse Events | |
| 8.3.1 | Time Period and Frequency for Collecting Adverse Event and Serious Adverse Information | |
| 8.3.2 | Method of Detecting Adverse Events and Serious Adverse Events | |
| 8.3.3 | Follow-up of Adverse Events and Serious Adverse Events | |
| 8.3.4 | Regulatory Reporting Requirements for Serious Adverse Events | |
| 8.3.5 | Pregnancy | |
| 0.5.5 | Tieghandy | 12 |
| 8.3.7 | Medication Errors | 43 |
| 8.4 | Treatment of Overdose | |
| 8.5 | Pharmacokinetics | |
| 8.6 | Pharmacodynamics | |
| 8.7 | Genetics | 44 |
| 8.9 | Medical Resource Utilization and Health Economics | 45 |
| 9. | Statistical Considerations | 46 |

| 9.1 | Statistical Hypotheses | 46 |
|---|---|---|
| 9.2 | Sample Size Determination | |
| 9.3 | Populations for Analyses | |
| 9.4<br>9.4.1 | Statistical Analyses | |
| | Efficacy Analyses | |
| | 4.1.1 Primary Efficacy Endpoints | |
| | 4.1.2 Primary Analyses | |
| | 4.1.3 Secondary Efficacy Endpoints | |
| | 4.1.4 Secondary Analyses | |
| | 4.1.5 Exploratory Efficacy Endpoints | |
| | 4.1.6 Exploratory Efficacy Analyses | |
| 9.4.2 | Safety Analyses | |
| | 4.2.1 Adverse Events | |
| | 4.2.2 Vital Signs | |
| | 4.2.3 Electrocardiograms | |
| 9.4.3 | , and the second se | |
| | 4.3.1 Immunogenicity Analyses | |
| 9.5 | Interim Analyses | |
| 10. | Supporting Documentation and Operational Considerations | 55 |
| 10.1 | Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | |
| 10.1.1 | Regulatory and Ethical Considerations. | |
| 10.1.2 | Financial Disclosure. | |
| 10.1.3 | Informed Consent Process | |
| 10.1.4 | Data Protection. | |
| 10.1.5 | Posting Clinical Study Data | |
| 10.1.6 | Data Quality Assurance | |
| 10.1.7 | Source Documents | |
| 10.1.8 | Study and Site Closure | 58 |
| 10.1.10 | 1 | |
| 10.2 | Appendix 2: Clinical Laboratory Tests | |
| 10.3 | Appendix 3: Adverse Events: Definitions and Procedures for Recording Follow-up, and Reporting | |
| Definitio | ion of AE | |
| | ion of SAE | |
| | ing and Follow-Up of AEs and/or SAEs | |
| | ing of SAEs | |
| 1 | <u> </u> | |



## **List of Figures**

## 1. Protocol Summary

## 1.1 Synopsis

**Protocol Title**: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of MT10109L (NivobotulinumtoxinA) for the Treatment of Glabellar Lines

**Protocol Number: MT10109L-001** 

**Brief Title**: MT10109L in the Treatment of Glabellar Lines

**Study Phase**: 3 **Study Rationale**:

The purpose of this placebo-controlled pivotal study is to evaluate the safety and efficacy of MT10109L for the treatment of glabellar lines (GL) in participants with moderate to severe GL

### **Objectives and Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary • To compare the efficacy between 20 U MT10109L and placebo for the treatment of GL in participants with moderate to severe GL | <ul> <li>For US FDA:</li> <li>Composite: The proportion of participants with a ≥ 2-grade improvement from baseline on the Facial Wrinkle Scale With Photonumeric Guide (FWS) according to investigator and participant assessments of GL severity at maximum frown at Day 30 using the intent-to-treat (ITT) population after a single intramuscular (IM) injection of MT10109L or placebo in the GL For EU regulatory agencies:</li> </ul> |
| <ul> <li>To compare the efficacy between MT10109L and placebo for the treatment of GL in participants with moderate to severe GL</li> <li>To compare the safety between MT10109L and placebo for the treatment of GL in participants with moderate to severe GL</li> </ul> | <ul> <li>Secondary: The duration of GL treatment effect, estimated as the median time to return to <i>moderate</i> or <i>severe</i> GL at maximum frown, in participants who achieved a rating of ≥ 2-grade improvement from baseline in GL severity at maximum frown at Day 30 according to investigator assessments using the FWS</li> <li>Secondary: The proportion of responders for investigator assessments of GL severity at maximum frown using the FWS, where a responder is defined as achieving a ≥ 2-grade improvement from baseline at maximum frown at Day 30</li> </ul> |



### **Overall Study Design:**

- This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 3 study to evaluate the safety and efficacy of MT10109L in treating GL.
- Participants are adults ≥ 18 years of age with moderate to severe GL at maximum frown (assessed by both the investigator and participant using the FWS [investigator and participant ratings must be the same for GL]).
- The primary efficacy measure is the investigators' and participants' assessments of GL at maximum frown using the FWS, and the primary timepoint is Day 30 after the first intervention.
- Participants will attend a Screening Visit up to 28 days before enrollment on Day 1.
- The first treatment period (Day 1 with follow-up to Day 180) is a double-blind, randomized, placebo-controlled, parallel-group, single treatment administration with a 6-month follow-up.
- On Day 1, participants will be randomly assigned in a 2:1 ratio to receive MT10109L 20 U or placebo.
- Participants who complete the study will have an exit visit at Day 360.

### **Number of Participants:**

Approximately 225 participants will be enrolled in order to have approximately 190 participants complete the study

### **Number of Sites:**

Approximately 16 global sites

### **Intervention Groups and Study Duration:**

- The total duration of study participation for each participant is approximately 12 months (Day 1 randomization/treatment to end of study/Day 360). Participants will attend the following visits:
  - o Screening (up to 28 days prior to Day 1)
  - o Randomization and treatment (Day 1)
  - o Follow-up visits on Days 7 and 14 after each intervention
  - o Monthly (Days 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, and 330)
  - o Exit (Day 360 [completion] or early exit)
- On Day 1, participants will receive IM injections of MT10109L 20 U or placebo.
- During the retreatment period (Day 180 through Day 330), participants who meet retreatment criteria will receive up to 2 open-label interventions of MT10109L 20 U

  Participants who complete the study will have an exit visit at Day 360.

**Data Monitoring Committee:** No









### 2. Introduction

### 2.1 Study Rationale

The purpose of this placebo-controlled, pivotal study is to evaluate the safety and efficacy of MT10109L for the treatment of GL in participants with moderate to severe GL

## 2.2 Background



Glabellar lines are deep furrows or *frown lines* in the glabellar area of the face, and LCL (or CFL) are horizontal *smile lines* by the sides of the eyes. Both types of facial lines result from the repetitive functional action of the underlying mimetic facial musculature during animation (Blitzer 1993). When injected at therapeutic doses, MT10109L produces partial chemical denervation of the muscle, resulting in localized reduction in muscle activity. Because GL and LCL result from muscular activity, the muscle relaxation leads to a temporary relief of facial lines. While it was previously thought that these facial lines were structural and permanent, the effects of these injections demonstrate the lines are part functional and remain because of constant muscle tone (Ferreira 2004; Garcia 1996).

The development of facial lines (such as GL and LCL) is an age-related change of the face that occurs because of the repetitive muscle contractions that are associated with common facial expressions. Thus, these facial lines can be observed with contraction (dynamic rhytides) or in more severe cases in repose (static rhytides). Increasing severity in the appearance of facial lines has been associated with a patient's perception of reduced attractiveness and a negative effect on self-esteem and sense of well-being (Koblenzer 1996). Furthermore, the appearance of these facial lines can lead to a miscommunication of an emotional state of anger, anxiety, disapproval, or sadness (Khan 2001) causing distress and affecting social interactions (Finn 2003).

Evidence supports that unattractive or aging skin is indeed related to psychological and psychosocial impacts (Farage 2010).

The popularity of BoNT/A cosmetic treatment of GL and LCL in adults is related to its proven efficacy for reducing moderate to severe facial lines (Beer 2006); well documented safety profile (Brin 2009); and positive impact on psychological well-being and the resulting psychosocial benefits (Finn 2003).



### 2.3 Benefit/Risk Assessment

Generally, the popularity of BoNT/A cosmetic treatment of GL and LCL in adults is related to its proven efficacy for reducing moderate to severe facial lines (Beer 2006); well documented safety profile (Brin 2009); and positive impact on psychological well-being and the resulting psychosocial benefits (Finn 2003). Compared with the general class of BoNT/A treatments, MT10109L provides additional benefits. For one, it is provided as a ready-to-use liquid product. Secondly, it is manufactured without human- or animal-derived products. MT10109L also offers

potential efficacy and safety advantages in addition to convenience since it does not require reconstitution and has shown sustained benefit in the treatment of GL.



## 3. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | For US FDA: |
| To compare the efficacy between 20 U MT10109L and placebo for the treatment of GL in participants with moderate to severe GL | <ul> <li>Composite: The proportion of participants with a ≥ 2-grade improvement from baseline on the FWS according to investigator and participant assessments of GL severity at maximum frown at Day 30 using the ITT population after a single IM injection of MT10109L or placebo in the GL For EU regulatory agencies:</li> <li>Coprimary: The proportion of participants achieving a rating of</li> </ul> |
| Secondary | For US FDA: |
| <ul> <li>To compare the efficacy between MT10109L and placebo for the treatment of GL in participants with moderate to severe GL</li> <li>To compare the safety between MT10109L and placebo for the treatment of GL in participants with moderate to severe GL</li> </ul> | <ul> <li>Secondary: The duration of GL treatment effect, estimated as the median time to return to moderate or severe GL at maximum frown, in participants who achieved a rating of ≥ 2-grade improvement from baseline in GL severity at maximum frown at Day 30 according to investigator assessments using the FWS</li> <li>Secondary: The proportion of responders for investigator assessments of GL severity at maximum frown using the FWS, where a responder is defined as achieving a ≥ 2-grade improvement from baseline at maximum frown at Day 30</li> <li>Secondary: The proportion of participants reporting mostly satisfied/very satisfied on the FLSQ follow-up version Item 5 for GL at Day 60</li> <li>Secondary: The proportion of responders for investigator assessments of GL severity at rest using the FWS among participants who were rated at least mild at rest at baseline, where a responder is defined as achieving a ≥ 1-grade improvement from baseline at Day 30</li> <li>Secondary: Incidence of adverse events; change from baseline in vital sign and ECG parameters; and presence of binding and neutralizing antibodies</li> <li>For EU regulatory agencies:</li> </ul> |





## 4. Study Design

### 4.1 Overall Design

- This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 3 study conducted across approximately 16 global sites to evaluate the safety and efficacy of MT10109L in treating GL. Participants may receive up to 3 study interventions (a single double-blind intervention of MT10109L 20 U or placebo and up to 2 open-label interventions with MT10109L 20 U).
- Participants are adults ≥ 18 years of age with moderate to severe GL at maximum frown (assessed by both the investigator and participant using the FWS [investigator and participant ratings must be the same for GL]).
- The primary efficacy measure is the investigators' and participants' assessments of GL severity at maximum frown using the FWS, and the primary timepoint is Day 30 after the first intervention.
- Participants will attend a Screening Visit up to 28 days before enrollment on Day 1.
- The first treatment period (Day 1 with follow-up to at least Day 180) is a double-blind, randomized, placebo-controlled, parallel-group, single treatment administration with a 6-month follow-up.
- On Day 1, participants will be randomly assigned in a 2:1 ratio to receive MT10109L 20 U or placebo.
- MT10109L 20 U or placebo will be administered as 5 IM injections: 5 to the GL complex (2 in each corrugator muscle, 1 in the procerus muscle), 0.1 mL (4 U MT10109L or 0 U placebo) per injection.
- Participants who complete the study will have an exit visit at Day 360.

- The total duration of study participation for each participant is approximately 12 months (Day 1 randomization/treatment to end of study/Day 360). Participants will attend the following visits:
  - o Screening (up to 28 days prior to Day 1)
  - o Randomization and treatment (Day 1)
  - o Follow-up visits on Days 7 and 14 after each intervention
  - Monthly (Days 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, and 330)
  - o Exit (Day 360 [completion] or early exit)



- Approximately 225 participants will be enrolled at approximately 16 global sites in order to have approximately 190 participants complete the study
- Participants who prematurely discontinue from the study will not be replaced.

#### 4.1.1 **Clinical Hypotheses**

MT10109L 20 U is more effective than placebo in treating GL, measured by both investigators' and participants' assessments of GL severity at maximum frown using the FWS.

MT10109L 20 U has an acceptable safety profile after single and repeat treatments.



## 4.4 End of Study Definition

The end of the study is defined as the date of the last scheduled procedure shown in the SoA for the last participant in the study globally.

A participant is considered to have completed the study if he/she has completed all phases of the study including the last scheduled procedure shown in the SoA.

## 5. Study Population

Participants in the current study have moderate to severe GL at maximum frown, as specified in Section 5.1.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

## 5.1 Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

| 1. | Age |
|---|---|
| 1.01 | Participant must be $\geq$ 18 years of age and considered to be an adult in her/his local jurisdiction at the time of signing the informed consent. |
| 2. | Type of Participant and Characteristics |
| 2.01 | Moderate to severe GL at maximum frown (as assessed by both the investigator and participant; ) using the FWS |
| 2.02 | Participants must have sufficient visual acuity without the use of eyeglasses (contact lens use acceptable) to accurately assess their GL lines, in the opinion of the investigator. |
| 3. | Sex |
| 3.01 | Male and female |
| 4. | Contraceptives |
| 4.01 | Female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period |
| 4.02 | Female participants of childbearing potential must have a negative urine pregnancy test before each study intervention. A female is considered NOT to be of childbearing potential if she is premenarchal, postmenopausal (at least 12 consecutive months without menstruation), or permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral oophorectomy). |

| 5. | Informed Consent |
|---|---|
| 5.01 | Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol |
| 5.02 | Written informed consent from the participant has been obtained prior to any study-related procedures. |



## 5.2

**5.2** Exclusion Criteria
Participants are excluded from the study if any of the following criteria apply:

| 1. | Medical Conditions |
|---|---|
| 1.01 | Any condition which precludes a participant's ability to comply with study requirements, including completion of the study visits or inability to read, understand, and/or self-assess GL severity using the FWS |
| 1.03 | Any medical condition that may put the participant at increased risk with exposure to MT10109L including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function |



| 2.06 | Prior facial treatment with permanent soft tissue fillers, synthetic implantation (eg, Gore-Tex®), and/or autologous fat transplantation |
|---|---|
| 3. | Prior/Concurrent Clinical Study Experience |
| 3.01 | Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study |
| 4. | Other |
| 4.01 | Females who are pregnant, nursing, or planning a pregnancy during the study |
| 4.02 | Participants who plan for an extended absence away from the immediate area of the study site that would preclude them from returning for all protocol specified study visits |



## **5.3** Lifestyle Considerations

No restrictions are required.



### 5.4 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the CONSORT publishing requirements and to respond to queries from health authorities. Minimal information includes demographics, screen failure details, eligibility criteria, and any SAE.

Screen failures can occur during the screening period up to the Day 1 Visit.

## 6. Study Intervention

Study intervention is defined as any investigational intervention(s), marketed product(s), or placebo intended to be administered to a study participant according to the study protocol.





### 6.1.2 Instructions for Use and Administration

Only trained and medically qualified physicians experienced with BoNT/A injections are authorized to administer the study interventions. Study-specific training for GL injections are provided to investigators

The GL study interventions will be administered as IM injections at 5 injection sites in the glabellar complex, 2 in each corrugator muscle and 1 in the procerus

Participants must be observed for adverse events for  $\geq 30$  minutes after each study intervention.



## 6.2 Preparation/Handling/Storage/Accountability

- 1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received and any discrepancies are reported and resolved before use of the study intervention.
- 2. Only participants enrolled in the study may receive study intervention, and only authorized site personnel may administer study intervention. All study intervention must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site personnel.

- 3. The investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (ie, receipt, reconciliation, and final disposition records).
- 4. Further guidance and information for the final disposition of unused study interventions are provided in the study manual.

All unused study intervention and empty vials must be returned to the sponsor at the termination of the study. Unit counts will be performed when the study intervention is returned, and all study intervention must be accounted for. Unused drug supplies and empty vials will be returned to the sponsor.



## **6.4** Study Intervention Compliance

Participants will receive all doses under the direct supervision of study site personnel. Study intervention compliance will not be calculated.

The study site will keep an accurate drug disposition record that specifies the amount of study intervention administered to each participant and the date of administration.

## 6.5 Concomitant Therapy

The use of any concomitant medication or vaccine (including prescription or over-the-counter medication, vitamins, and/or herbal supplements) is to be recorded on the participant's eCRF at each visit along with the reason the medication is taken.

At screening and end of study and upon admission to and discharge from the study site, study site personnel will question each participant specifically on the use of concomitant medications. Study site personnel must notify the sponsor immediately if a participant consumes any concomitant medications not permitted by the protocol. Participants who admit to using prohibited concomitant medications may be discontinued from the study at the discretion of the investigator or the sponsor.





### 6.5.3 Rescue Medicine

Rescue medicine is not applicable.

## **6.6** Dose Modification

This protocol does not allow for alteration from the currently outlined dosing schedule.





Approval Date: 30-Sep-2020 22:56:38 (GMT)

### 7. **Discontinuation of Study Intervention and Participant** Discontinuation/Withdrawal

A premature discontinuation will occur if a participant who signs the ICF and is randomized ceases participation in the study, regardless of circumstances, before the completion of the protocol-defined study procedures.

Notification of early participant discontinuation from the study and the reason for discontinuation will be made to the sponsor and will be clearly documented on the appropriate eCRF.

Reasons for discontinuation from the study intervention and/or the study may include the following commonly used terms:

| Commonly Used Terms |
|-----------------------------|
| Adverse event |
| Lost to follow-up |
| Lack of efficacy |
| Other |
| Physician decision |
| Pregnancy |
| Protocol deviation |
| Site terminated by sponsor |
| Study terminated by sponsor |
| Withdrawal by subject |

#### 7.1 **Discontinuation of Study Intervention**

Study intervention should be discontinued for the following reasons:

- Pregnancy
- Other safety criteria

Women who test positive for urine pregnancy test will NOT receive further treatment and will be discontinued from the study. They should complete study exit procedures and be followed up for pregnancy outcome. See the SoA for data to be collected at the time of intervention discontinuation and follow-up and for any further evaluations that need to be completed.

## 7.2 Participant Discontinuation/Withdrawal from the Study

- A participant may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons.
- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- See the SoA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.

## 7.3 Lost to Follow Up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the study site for a required study visit:

- The study site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make
  every effort to regain contact with the participant (where possible, 3 telephone calls and,
  if necessary, a certified letter to the participant's last known mailing address or local
  equivalent methods). These contact attempts will be documented in the participant's
  medical record.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

## 8. Study Assessments and Procedures

- Study procedures and their timing are summarized in the SoA.
- Immediate safety concerns should be discussed with the sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.
- Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.



## 8.1 Efficacy Assessments

## 8.1.1 Facial Wrinkle Scale With Photonumeric Guide (FWS)

Investigators' and participants' assessments of the severity of GL at rest and maximum frown using the validated FWS, based on the following scale:

- 0 = None
- 1 = Mild
- 2 = Moderate
- 3 = Severe






## 8.2 Safety Assessments

Planned timepoints for all safety assessments are provided in the SoA.

## **8.2.1** Adverse Events

The investigator will question the participant to ascertain whether any adverse events were experienced since the previous visit. Additionally, at treatment visits, the participants will be observed for  $\geq 30$  minutes following study intervention. All pertinent information regarding adverse events (ie, date of onset and stop, duration, outcome, severity, relationship to study intervention, action or treatment required) will be obtained and recorded in the source documents and appropriate eCRF page.

## 8.2.2 Physical Examination





## 8.2.4 Vital Signs

Pulse rate (beats per minute): Participants are to be seated for at least 2 minutes, and pulse rate will be counted over 60 seconds, and recorded in the source document and eCRF as beats per minute.

Blood pressure (mm Hg): Participants are to be seated for at least 2 minutes, and systolic/diastolic blood pressure will be measured.

Respiration rate (breaths per minute): Participants are to be seated for at least 2 minutes, and breaths will be counted for 30 seconds and multiplied by 2.

## 8.2.5 Electrocardiograms

- All participants will undergo conventional 12-lead ECG using standardized equipment and
  electrode placement at the visits outlined in the SoA. Participants are to be in a
  semirecumbent position for at least 10 minutes prior to starting the tracing. During screening,
  a single ECG trace will be taken to assess entry eligibility.
- A qualified third-party vendor will read the ECGs and report the findings as normal, abnormal, or unable to evaluate.



• The ECG will be assessed for the following measures: heart rate, QRS duration, QT interval, QTcB interval, QTcF interval, ST segment, RR interval, PR interval, and qualitative results.

## 8.2.6 Hematology and Blood Chemistry

- See Appendix 2 for the list of clinical laboratory tests to be performed and the SoA for the timing and frequency.
- Hematology and nonfasting blood chemistry assays will be performed by a central laboratory.
- During the Screening Period, the investigator or subinvestigator will assess the clinical significance of any values outside the reference ranges provided by the laboratory, and participants with abnormalities judged to be clinically significant will be excluded from the study.

## 8.2.7 Urine Pregnancy Tests

Urine dipstick kits will be used to conduct pregnancy tests at the timepoints specified in the SoA, or more frequently, at the investigator's discretion.

## 8.2.8 Suicidal Risk Monitoring

Suicidal risk monitoring is not applicable for this study.

## 8.3 Adverse Events and Serious Adverse Events

The definitions of an adverse event or SAE can be found in Appendix 3.

Adverse events will be reported by the participant.

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an adverse event or SAE and remain responsible for following up adverse events that are serious, considered related to the study intervention or study procedures, or that caused the participant to discontinue the study intervention (see Section 7).

Adverse drug reactions for MT10109L have not been established.

The following expected adverse drug reactions are based on BOTOX clinical trial data for the treatment of GL (Table 8-1).

Table 8-1 Expected Adverse Reactions for Treatment of Glabellar Lines

| Expected Adverse Reactions <sup>a</sup> | Incidence |
|-----------------------------------------|-----------|
| Eyelid ptosis | 3% |
| Facial pain | 1% |
| Facial paresis | 1% |
| Muscular weakness | 1% |

<sup>&</sup>lt;sup>a</sup> Data are based on BOTOX glabellar lines clinical trial data (BOTOX Cosmetic US Package Insert, 2017)

The adverse drug reactions of eyelid ptosis, facial pain, facial paresis, and muscular weakness usually are mild in severity, reversible, and have a low incidence. Therefore, no treatment for these reactions is recommended. If these reactions are moderate or severe, medical help should be sought as needed.

# 8.3.1 Time Period and Frequency for Collecting Adverse Event and Serious Adverse Event Information

For participants who received study intervention, all adverse events from the signing of the ICF until 30 days after the last study visit will be collected at the timepoints specified in the SoA and as observed or reported spontaneously by study participants.

Medical occurrences that begin before the start of study intervention, but after obtaining informed consent will be recorded in the adverse event section of the eCRF.

All SAEs from the signing of the ICF until at least 12 weeks after the last administration of study intervention will be collected at the timepoints specified in the SoA (Section 1.3), and as observed or reported spontaneously by study participants.

All SAEs will be recorded and reported to the sponsor or designee within 24 hours, as indicated in Appendix 3. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek adverse event or SAE information after conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify the sponsor.

The method of recording, evaluating, and assessing causality of adverse events and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3.

## 8.3.2 Method of Detecting Adverse Events and Serious Adverse Events

Care will be taken not to introduce bias when detecting adverse events and/or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about adverse event occurrences.

## 8.3.3 Follow-up of Adverse Events and Serious Adverse Events

| After the initial adverse event/SAI | E report, the investigator is required to proactively follow each |
|---|---|
| participant who received study int | ervention at subsequent visits/contacts. All TEAEs/SAEs, |
| including AESIs | will be followed until resolution, stabilization, the event is |
| otherwise explained, or the partici | pant is lost to follow-up |

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the sponsor to elucidate the nature and/or causality of the adverse event or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide the sponsor with a copy of any postmortem findings including histopathology.

New or updated information will be recorded in the originally completed eCRF.

The investigator will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

## **8.3.4** Regulatory Reporting Requirements for Serious Adverse Events

- Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.
- The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRBs/ IECs, and investigators.
- Investigator safety reports must be prepared for SUSARs according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.
- An investigator who receives an investigator safety report describing an SAE or other specific safety information (eg, summary or listing of SAEs) from the sponsor will review and then file it along with the investigator's brochure and will notify the IRB/IEC, if appropriate according to local requirements.

## 8.3.5 Pregnancy

- Urine pregnancy testing will be conducted for women of childbearing potential prior to each study intervention, and at the study exit visit. See Appendix 7 for detailed information on definition of women of childbearing potential, use of contraceptives, and pregnancy.
- To minimize the risk of pregnancy, all women of childbearing potential must agree to use a highly effective or acceptable contraception method (Appendix 7) consistently and correctly throughout the duration of the study.
- Women who test positive for urine pregnancy test will NOT receive further treatment and will be discontinued from the study.
- Women who test positive for urine pregnancy test should complete end-of-study procedures and be followed up for pregnancy outcome.

- Any termination of pregnancy will be reported, regardless of fetal status (presence or absence of anomalies) or indication for the procedure.
- If a pregnancy is reported, the investigator should inform the sponsor within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 7.
- Abnormal pregnancy outcomes (eg, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) or genetic abnormalities (whether leading to an elective abortion or not) are considered SAEs.

## 8.3.7 Medication Errors

Medication error refers to any unintended error in the dosing and/or administration of the study intervention as per instructions in the protocol. Medication errors generally fall into 4 categories as follows:

- Wrong study intervention
- Wrong dose (including dosing regimen, strength, form, concentration, amount)
- Wrong route of administration
- Wrong participant (ie, not administered to the intended participant)

Medication errors include occurrences of overdose and underdose of the study intervention.

Overdose: Unintentional administration of a quantity of the study intervention given per administration that is above the maximum recommended dose according to the protocol for the study intervention or comparator as applicable. See Section 8.4 for information on the treatment of overdose.

Underdose: Unintentional administration of a quantity of the study intervention given per administration that is under the minimum recommended dose according to the protocol.

## **8.4** Treatment of Overdose

Overdose of MT10109L is a relative term and depends upon dose, site of injection, and underlying tissue properties. Signs and symptoms of overdose are likely not to be apparent immediately postinjection. Excessive doses may produce local, or distant, generalized and profound neuromuscular paralysis.

Because MT10109L is administered as injections by physicians, for this study, the chance of overdose is extremely low. Should accidental injection or oral ingestion occur or overdose be suspected, the participant should be medically monitored for up to several weeks for progressive

signs or symptoms of systemic muscular weakness that could be local or distant from the site of injection, which may include ptosis, diplopia, dysphagia, dysarthria, generalized weakness, or respiratory failure. For GL or LCL, eyelid ptosis, diplopia, and vision blurred are known local effects of the toxin. These participants should be considered for further medical evaluation and appropriate medical therapy immediately instituted, which may include hospitalization.

If the musculature of the oropharynx and esophagus is affected, aspiration may occur, which may lead to development of aspiration pneumonia. If the respiratory muscles become paralyzed or sufficiently weakened, intubation and assisted respiration may be necessary until recovery takes place. Supportive care could involve the need for a tracheostomy and/or prolonged mechanical ventilation, in addition to other general supportive care.

In the event of an overdose, the investigator should educate the participant, monitor the course of overdose, contact the medical safety physician as needed, document the quantity of the excess dose, associated adverse events as well as the duration of the overdose in the eCRF.

## 8.5 Pharmacokinetics

Pharmacokinetic parameters are not evaluated in this study.

## 8.6 Pharmacodynamics

Pharmacodynamic parameters are not evaluated in this study.

## 8.7 Genetics

Genetics are not evaluated in this study.





## **8.9** Medical Resource Utilization and Health Economics

Medical resource utilization and health economics parameters are not evaluated in this study.

## 9. Statistical Considerations

## 9.1 Statistical Hypotheses

For US FDA:

The primary efficacy analysis will be performed on the ITT population, which consists of all randomized participants. The following hypotheses will be used to compare MT10109L 20 U with placebo:

- Null hypothesis: MT10109L 20 U and placebo are equally effective in reducing GL severity at maximum frown as measured by the proportion of responders with a ≥ 2-grade improvement from baseline based on both the investigator- and participant-rated FWS at Day 30.
- Alternative hypothesis: MT10109L 20 U and placebo are not equally effective in reducing GL severity at maximum frown as measured by the proportion of responders with a ≥ 2-grade improvement from baseline based on both the investigator- and participant-rated FWS at Day 30.

For EU regulatory agencies:



## 9.2 Sample Size Determination

Approximately 225 participants will be randomized into the study in a 2:1 ratio yielding approximately 150 participants in the MT10109L 20 U group and 75 participants in the placebo group in the first treatment period. The sample size of 225 allows for an adequate safety database of participants treated with MT10109L for this indication.



## 9.3 Populations for Analyses

Primary and secondary efficacy analyses for the US FDA will be performed on the ITT population, consisting of all randomized participants.



The safety analyses will be based on the safety population, which will include all participants who receive at least 1 injection of study intervention. All safety analyses will be performed with participants analyzed by their actual treatment or regimen received.

## 9.4 Statistical Analyses

The SAP will be developed and finalized before database lock and unblinding and will describe the participant populations to be included in the analyses, and procedures for accounting for missing, unused, and spurious data. This section is a summary of the planned statistical analyses of the primary, secondary, and exploratory endpoints.

## 9.4.1 Efficacy Analyses

## 9.4.1.1 Primary Efficacy Endpoints

For the US FDA, the composite efficacy endpoints are the proportion of participants with a  $\geq$  2-grade improvement from baseline on the FWS according to both investigator and participant assessments of GL severity at maximum frown at Day 30 using the ITT population after a single IM injection of MT10109L or placebo in the GL.

## 9.4.1.2 Primary Analyses

The primary efficacy analysis will be based on the comparison of GL efficacy for MT10109L 20 U versus placebo at the primary timepoint of Day 30 of the first treatment period. The evaluation of the equality of the proportions of responders will be based on CMH test stratified by investigator-assessed baseline GL severity at maximum frown. Relative risk and 95% CI for relative risk will be presented. Missing values will be imputed up to Day 180 using multiple imputation methods. SAS Proc MI procedure will be used

| Seed for all Proc MI procedure is prespecified as |
|---------------------------------------------------|





The primary efficacy variables will be evaluated across all study visits, with the primary timepoint being Day 30 of the first treatment period.

Sensitivity analyses of the primary efficacy variables will be performed to establish their consistency and robustness as well as to further characterize the extent of participants' responses.

## 9.4.1.3 Secondary Efficacy Endpoints

For US FDA:

- The duration of GL treatment effect estimated as the median time to return to *moderate* or *severe* GL at maximum frown, in participants who achieved a rating of ≥ 2-grade improvement from baseline in GL severity at maximum frown at Day 30 according to investigator assessments using the FWS.
- The proportion of responders for investigator assessments of GL severity at maximum frown using the FWS, where a responder is defined as achieving a  $\geq$  2-grade improvement from baseline at maximum frown at Day 30



- The proportion of participants reporting *mostly satisfied/very satisfied* on the FLSQ follow-up version Item 5 for GL at Day 60.
- The proportion of responders for investigator assessments of GL severity at rest using the FWS, among participants who were rated at least *mild* at rest at baseline, where a responder is defined as achieving a  $\geq$  1-grade improvement from baseline at Day 30.

For EU regulatory agencies:





## 9.4.1.4 Secondary Analyses

All secondary variables will be evaluated for all study visits with the prespecified primary timepoint given above, except for duration of treatment effect. The duration of GL treatment effect is defined as the time to return to moderate or severe GL at maximum frown, in those participants achieving a responder status (for US FDA, responder is defined as participants who achieved a rating of  $\geq$  2-grade improvement from baseline in GL severity at maximum frown;

at Day 30 according to investigator assessments using the FWS. It will be estimated using the Kaplan-Meier method.

A serial gatekeeping strategy will be used to account for multiplicity in testing the primary and secondary efficacy variables at the primary timepoint

The proportion of responders will be analyzed using the CMH test stratified by baseline GL severity at maximum frown as assessed by the clinician (investigator or subinvestigator). The continuous variables and ordinal variables will be analyzed using ANCOVA

## 9.4.1.5 Exploratory Efficacy Endpoints

For both the US FDA and EU, analyses for exploratory efficacy endpoints will be performed on the ITT population.



The proportion of responders will be analyzed using the CMH test

## 9.4.2 Safety Analyses

The safety analysis will be performed using the safety population and are fully defined in the SAP. The safety parameters will include:

| • | Adverse events |
|---|----------------|

- Vital signs
- Electrocardiogram
- Immunogenicity analyses

## 9.4.2.1 Adverse Events

An adverse event will be considered a TEAE if:

- The adverse event began on or after the date of the first dose of study intervention; or
- The adverse event was present before the date of the first dose of study intervention, but increased in severity or became serious on or after the date of the first dose of study intervention

An adverse event that occurs more than 30 days after study exit will not be counted as a TEAE.

An adverse event will be considered a TESAE if it is a TEAE that additionally meets any SAE criteria.

The number and percentage of participants reporting TEAEs in each study intervention group will be tabulated by system organ class and preferred term and by system organ class, preferred term, and severity.

The number and percentage of participants reporting treatment related TEAEs in each study intervention group will be tabulated by system organ class and preferred term.

The number and percentage of participants reporting TEAEs that are included in the PDSOT <u>term list</u> will be tabulated by study intervention group.

Summary tables will be provided for participants with SAEs and participants with adverse events leading to discontinuation if 5 or more participants reported such events. Listings of all adverse events, SAEs, and adverse events leading to discontinuation by participant will be presented.

The definitions of an adverse event and SAE can be found in Appendix 3.

## 9.4.2.2 Vital Signs

Descriptive summaries (n, mean, SD, median, minimum, and maximum) of actual values and changes from baseline will be calculated for vital signs (systolic and diastolic blood pressure, pulse and respiration rate). These summaries will be presented by study intervention and by visit.

## 9.4.2.3 Electrocardiograms

Descriptive statistics for ECG parameters (eg, heart rate, QRS duration, QT interval, QTc intervals, RR interval, and PR interval) at baseline, and changes from baseline at all postbaseline timepoints will be presented by study intervention and by visit. For each parameter, only participants who had both baseline postbaseline assessments will be included in the summary.

## 9.4.3 Other Analyses

## 9.4.3.1 Immunogenicity Analyses

Immunogenicity results, manifested as the presence of binding antibodies and neutralizing antibodies to MT10109L, will be summarized in a table.

## 9.5 Interim Analyses

No interim analysis is planned.

## 10. Supporting Documentation and Operational Considerations

# 10.1 Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

## 10.1.1 Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with the following:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
  - o Applicable ICH/ISO GCP guidelines
  - Applicable laws and regulations
- The protocol, protocol amendments, ICF, investigator's brochure, and other relevant documents (eg, advertisements) must be submitted to an IRB/IEC by the investigator and reviewed and approved by the IRB/IEC before the study is initiated.
- Any amendments to the protocol will require IRB/IEC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
  - Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
  - o Providing oversight of the overall conduct of the study at the site and adherence to requirements of applicable local regulations, for example 21 CFR, ICH guidelines, the IRB/IEC, and European regulation 536/2014 for clinical studies (if applicable)

## **10.1.2** Financial Disclosure

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.



## 10.1.3 Informed Consent Process

- The investigator or his/her representative will explain the nature of the study to the participant or his/her legally authorized representative and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, HIPAA requirements, where applicable, and the IRB/IEC or study center.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be reconsented to the most current version of the ICF(s) during their participation in the study.
- A copy of the ICF(s) must be provided to the participant or the participant's legally authorized representative.

Participants who are rescreened are required to sign a new ICF.

#### 10.1.4 Data Protection

- Participants will be assigned a unique identifier. Any participant records or datasets that are transferred to the sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.
- The participant must be informed that his/her medical records may be examined by clinical quality assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

## 10.1.5 Posting Clinical Study Data

- Clinical study reports, safety updates, and annual reports will be provided to regulatory authorities as required.
- Company-sponsored study information and tabular study results will be posted on the US National Institutes of Health's website www.ClinicalTrials.gov and other publicly accessible sites.

## **10.1.6** Data Quality Assurance

- All participant data relating to the study will be recorded on printed or eCRFs unless transmitted to the sponsor or designee electronically (eg, laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF.
- The investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- The sponsor or designee is responsible for the data management of this study including quality checking of the data.
- Study monitors will perform ongoing source data verification to confirm that data entered into the eCRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.
- Records and documents, including signed ICFs, pertaining to the conduct of this study must be retained by the investigator as stated in the clinical trial agreement. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor.

#### 10.1.7 Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.
- Data reported on the CRF or entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study.
- Definition of what constitutes source data can be found in Section 4.0 of ICH E6, Good Clinical Practice: Consolidated Guidance and must follow ALCOA, ie, records must be attributable, legible, contemporaneous, original, and accurate.

## 10.1.8 Study and Site Closure

The sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the investigator
- Discontinuation of further study intervention development



## **10.1.10** Compliance with Protocol

The investigator is responsible for compliance with the protocol at the investigational site and will ensure the availability of appropriate study personnel and compliance with GCP regulations and procedures. Trainings are provided by the sponsor to discuss the protocol procedures and study requirements. A representative of the sponsor will make frequent contact with the investigator and his/her research staff and will conduct regular monitoring visits at the site to review participant and study intervention accountability records for compliance with the protocol. Protocol deviations will be discussed with the investigator upon identification. The use of the data collected for the participant will be discussed to determine if the data are to be included in the analysis. The investigator will enter data that may be excluded from analysis as defined by the protocol deviation specifications. Significant protocol deviations will be reported to the IRB/IEC according to the IRB/IEC's reporting requirements.

# Approval Date: 30-Sep-2020 22:56:38 (GMT)

#### 10.2 **Appendix 2: Clinical Laboratory Tests**

- The tests detailed in Table 10-1 will be performed by the central laboratory.
- Protocol-specific requirements for inclusion or exclusion of participants are detailed in Section 5 of the protocol.
- Additional tests may be performed at any time during the study as determined necessary by the investigator or required by local regulations.

**Table 10-1 Protocol-required Safety Laboratory Assessments** 

| Laboratory<br>Assessments | | Parameters |
|---|---|---|
| Hematology | Platelets | WBC count with differential (absolute): |
| | RBC count | Neutrophils |
| | Hemoglobin | Lymphocytes |
| | Hematocrit | Monocytes |
| | RBC morphology | Eosinophils |
| | | Basophils |
| Clinical | BUN | Glucose |
| Chemistry | Potassium | Calcium |
| | AST | Alkaline phosphatase |
| | Total, direct, and indirect bilirubin | Chloride |
| | Creatinine | Albumin |
| | Sodium | Magnesium |
| | ALT | Phosphorus |
| | Total protein | Bicarbonate (carbon dioxide content) |
| | | Uric acid |

Investigators must document their review of each laboratory safety report.

# 10.3 Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

## **Definition of AE**

## **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.



## **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (eg, ECGs, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator (ie, not related to progression of underlying disease); for example:
  - o The test result is associated with accompanying symptoms, and/or
  - The test result requires additional diagnostic testing or medical/surgical intervention, and/or

- The test result leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy, and/or
- o The test result is considered to be an AE by the investigator or sponsor.
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition
- New condition detected or diagnosed after study intervention administration even though it may have been present before the start of the study
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE or SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.
- Lack of efficacy or failure of expected pharmacological action per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as AEs or SAEs if they fulfil the definition of an AE or SAE.

## **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety
  assessments that are associated with the underlying disease, unless judged by the
  investigator to be more severe than expected for the participant's condition. Merely
  repeating an abnormal test, in the absence of any of the above conditions, does not
  constitute an AE. Any abnormal test result that is determined to be an error does not
  require recording as an AE.
- The disease/disorder being studied or expected progression, signs, or symptoms (clearly defined) of the disease/disorder being studied, unless more severe than expected for the participant's condition
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital)

• Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen

#### **Definition of SAE**

SAEs must meet both the AE criteria described above and the seriousness criteria listed below.

## An SAE is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

## b. Is life threatening

The term *life threatening* in the definition of *serious* refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

## c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or intervention that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether hospitalization occurred or was necessary, the AE should be considered serious.

Hospitalization for elective intervention of a pre-existing condition that did not worsen from baseline is not considered an AE.

## d. Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

## e. Is a congenital anomaly/birth defect

## f. Other situations:

Medical or scientific judgment should be exercised in deciding whether SAE
reporting is appropriate in other situations such as important medical events that may
not be immediately life threatening or result in death or hospitalization but may
jeopardize the participant or may require medical or surgical intervention to prevent
one of the other outcomes listed in the above definition. These events should usually
be considered serious

Examples of such events include invasive or malignant cancers, intensive intervention in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

## Recording and Follow-Up of AEs and/or SAEs

## **AE and SAE Recording**

- When an AE or SAE occurs, it is the responsibility of the investigator to review all
  documentation (eg, hospital progress notes, laboratory reports, and diagnostics
  reports) related to the event.
- The investigator will then record all relevant AE or SAE information in the eCRF.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to the sponsor in lieu of completion of the AE or SAE eCRF page.
- There may be instances when copies of medical records for certain cases are requested by the sponsor. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to the sponsor.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.



| Assessment of | Intensity |
|---|---|
| MILD | A type of adverse event that is usually transient and may require only minimal |
| | treatment or therapeutic intervention. The event does not generally interfere |
| | with usual activities of daily living. |
| MODERATE | A type of adverse event that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. |
| SEVERE | A type of adverse event that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. |

An event is defined as *serious* when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

## **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE or SAE.
- A *reasonable possibility* of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other
  risk factors, as well as the temporal relationship of the event to study intervention
  administration will be considered and investigated.
- The investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE or SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE or SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor.



- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

## **Reporting of SAEs**

## **SAE Reporting**

• In rare circumstances and in the absence of facsimile equipment, notification by telephone is acceptable with a copy of the SAE form, sent by overnight mail or courier service.

• Initial notification via telephone does not replace the need for the investigator to complete and sign the SAE form within the designated reporting time frames.

## 10.4 Appendix 4: Abbreviations

| Term/Abbreviation | Definition |
|---|---|
| AESI | adverse event of special interest |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AST | aspartate aminotransferase |
| BoNT/A | botulinum toxin type A |
| BUN | blood urea nitrogen |
| CFL | crow's feet lines |
| CIOMS | Council for International Organizations of Medical Sciences |
| CMH | Cochran-Mantel-Haenszel |
| CONSORT | Consolidated Standards of Reporting Trials |
| CFR | Code of Federal Regulations |
| DVD | digital versatile disc |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| ELISA | enzyme-linked immunosorbent assay |
| EU | European Union |
| FDA | Food and Drug Administration |
| FLO-11 | 11-item Facial Line Outcomes questionnaire |
| FLSQ | Facial Line Satisfaction Questionnaire |
| FWS | Facial Wrinkle Scale with Photonumeric Guide |
| GCP | Good Clinical Practices |
| GL | glabellar lines |
| HIPAA | Health Insurance Portability and Accountability Act |
| IB | investigator's brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IM | intramuscular |
| IND | investigational new drug application |

IRB Institutional Review Board

ITT intent-to-treat

IUD intrauterine device

IWRS interactive web response system

LCL lateral canthal lines

LLN lower limit of normal value provided by the laboratory

mITT modified intent-to-treat

PRO patient-reported outcome

RBC red blood cells

SAE serious adverse event SAP statistical analysis plan

SI Le Système International d'Unités (International System of Units)

SoA schedule of activities
SUSAR serious adverse reactions

TCA trichloroacetic acid

TEAE treatment-emergent adverse events

U Units

UFL upper facial lines

ULN upper limit of normal value provided by the laboratory

US United States
WBC white blood cells














































## 10.10 Appendix 10: Protocol Amendment History

The protocol amendment summary of changes table for the current amendment is located directly before the table of contents.

### Amendment 1 (September 2018)

This amendment is considered to be nonsubstantial

The editorial nature of this amendment is intended to provide clarity of information throughout the document.

#### **Overall Rationale for the Amendment:**

The overall rationale for the changes implemented in the protocol amendment were administrative in nature.



### **Amendment 2 (November 2018)**

This amendment is considered to be nonsubstantial

# CONFIDENTIAL MT10109L

### **Overall Rationale for the Amendment:**

The overall rationale for the change implemented in the protocol was administrative in nature.

| Section No.<br>and Name | Description of Change | Brief Rationale |
|-------------------------|------------------------|-----------------|
| Title Page | Added Allergan Limited | Administrative |

## **Amendment 3 (February 2019)**

This amendment is considered to be substantial







## CONFIDENTIAL MT10109L

| Section No. and Name | Description of Change | Brief Rationale |
|---|---|---|
| 9.4.2.1 (Adverse Events) | Added a paragraph describing analysis of TEAEs related to possible distant spread of toxin (PDSOT) and monitoring of PDSOT | Clarification of process |
| 9.4.2.2 (Vital Signs) and 9.4.2.3 (Electrocardiograms) | Modified the description of analyses for clarity | Improve clarity |
| Appendix 1 (subsection of Compliance with Protocol) | Added text to clarify compliance with GCP regulations and procedures, and training of investigators on study requirements | Updated per recommendation by health authority |
| Appendix 7 | Revised criteria for postmenopausal females who are not being considered women of childbearing potential | Improve clarity |
| Appendix 7 (Table 10-2) | Added text to include as one of the acceptable birth control methods the option of male or female condoms without spermicide (in addition to male or female condoms with spermicide) | Correction |
| Throughout | Minor editorial revisions | Minor, therefore<br>have not been<br>summarized |

CONFIDENTIAL MT10109L

## 11. References

Beer KR. Comparative evaluation of the safety and efficacy of botulinum toxin type A and topical creams for treating moderate-to-severe glabellar rhytids. Dermatol Surg. 2006;32:184-192.

Blitzer A, Brin MF, Keen MS, Aviv JE. Botulinum toxin for the treatment of hyperfunctional lines of the face. Arch Otolaryngol Head Neck Surg. 1993;119:1018-1022.

BOTOX® Cosmetic (onabotulinumtoxinA) for injection [package insert]. Irvine, CA: Allergan, Inc; October 2017.

Brin MF, Boodhoo TI, Pogoda JM, James LM, Demos G, Terashima Y, et al. Safety and tolerability of onabotulinumtoxinA in the treatment of facial lines: A meta-analysis of individual patient data from global clinical registration studies in 1678 participants. J Am Acad Dermatol. 2009;61:961-970.e1-11.

Dmitrienko A, Molenberghs G, Chuang-Stein C, Offen W. Gatekeeping Strategies. In: Analysis of clinical trials using SAS: a practical guide. Cary, NC: SAS Institute; 2005. p. 104-108.

Farage MA, Miller KW, Berardesca E, Maibach HI. Psychological and Social Implications of Aging Skin: Normal Aging and the Effects of Cutaneous Disease. In: Farage MA, Miller KW, Maibach HI, editors. Textbook of Aging Skin. Springer; New York, New York: 2010;949-957.

Ferreira MC, Salles AG, Gimenez R, Soares MFD. Complications with the use of botulinum toxin type A in facial rejuvenation: report of 8 cases. Aesthet Plast Surg. 2004;28:441-444.

Finn CJ, Cox SE, Earl ML. Social implications of hyperfunctional facial lines. Dermatol Surg. 2003;29:450-455.

Garcia A, Fulton JE Jr. Cosmetic denervation of the muscles of facial expression with botulinum toxin: A dose-response study. Dermatol Surg. 1996;22:39-43.

Khan JA. Aesthetic surgery: Diagnosing and healing the miscues of human facial expression. Ophthal Plastic Reconstr Surg. 2001;17:4-6.

Koblenzer CS. Psychologic aspects of aging and the skin. Clin Dermatol. 1996;14:171-177.



O'Kelly M, Ratitch B. Clinical trials with missing data: A guide for practitioner. Statistics in Practice. Wiley; 2014.

Wilson EB, Hilferty, MM. The distribution of chi-squared. Proceedings of the National Academy of Sciences, Washington. 1931;17:12,684–688.

